CLINICAL TRIAL: NCT06509282
Title: Efficacy of a Personalized Concurrent Exercise Prescription Guide for Controlling Cardiovascular Risk and Enhancing Physical Fitness in Adults From a Cardiovascular Health Program: A Pilot Randomized Controlled Clinical Trial.
Brief Title: Personalized Concurrent Exercise for Cardiovascular Risk Control and Fitness in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Sebastián (Other)
Responsible Party: Principal Investigator, Johnattan Cano Montoya, Principal Investigator, Universidad San Sebastián
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5352023
Record Dates: First submitted 2024-05-24; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Syndrome, Metabolic
Keywords: Exercise; Concurrent training; Cardiovascular risk; Physical Fitness; Global rate scale; Adherence
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The concealment of allocation will be conducted by a researcher not involved in the clinical procedures of the intervention using the method of opaque, sealed, and consecutively numbered envelopes. The random sequence and allocation concealment allow for the control of selection bias.
  For enhanced bias control, the data analysis will be performed by a researcher blinded to the intervention groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concurrent training (Experimental): Concurrent training group
  Interventions: Behavioral: Concurrent training
- Control (No Intervention): Control group

INTERVENTIONS:
Behavioral: Concurrent training — Protocol:
  Duration: 6 weeks. Frequency: 3 times a week. Type: Concurrent. This consists of a combination of aerobic exercise and muscular resistance exercise.
  Details of the type of exercise:
  Aerobic exercise:
  Participants will perform 5-10 intervals per session of walking or jogging at a moderate to high intensity, with a rating of 5 to 10 points on the modified Borg scale of 1-10 points. Each interval will consist of 1 minute of walking or jogging, followed by 2 minutes of inactive pause.
  Muscular resistance exercise:
  Participants will perform concentric and eccentric and/or isometric contractions for 1 minute at an intensity of 5-10 according to the OMNI-RES scale. The rest period will last 2 minutes, and each exercise will be repeated 3 times. Three exercises per session will be performed: squats, push-ups, and plank.
  Pharmacological treatment:
  Participants will be asked to maintain their lifestyle, including taking prescribed medication as usual.
  Arms: Concurrent training

SUMMARY:
Aim: To determine the efficacy of a personalized concurrent exercise prescription guide combined with pharmacological treatment compared to pharmacological treatment alone in controlling cardiovascular risk factors and physical capacity in adults enrolled in a Cardiovascular Health Program.

Research Design: This pilot randomized controlled clinical trial (RCT) evaluates the efficacy of a personalized concurrent exercise prescription guide combined with pharmacological treatment versus pharmacological treatment alone. Outcomes: blood pressure, fasting glucose, total cholesterol, and triglycerides, muscle strength, cardiorespiratory capacity, body composition, adherence to the exercise guide, and patient perception of intervention effects, sociodemographic and medical background, physical activity level, Population: Adult users of the Cardiovascular Health Program at the External CESFAM in Valdivia will be recruited during regular check-up hours. Detailed study information will be provided, and informed consent obtained.

Sample Size: The sample size is 15 subjects per group, accounting for a 30% dropout rate, resulting in 39 participants. Participants will be randomly assigned to experimental (EG) or control groups (CG) with a 1:1 allocation ratio. Allocation concealment will be ensured with opaque, sealed envelopes.

Evaluations: Pre- and post-intervention evaluations will be conducted in both groups. Sociodemographic and medical background information will be collected through clinical record reviews. Blood pressure, heart rate, glucose, triglycerides, cholesterol, adherence to the exercise guide, and patient perception of intervention effects will be measured using standardized procedures by trained kinesiologists.

DETAILED DESCRIPTION:
SCIENTIFIC COMPONENT, METHODOLOGY, ETHICS, AND PLANNING

RESEARCH QUESTION AND HYPOTHESIS Research Question What is the efficacy of a personalized concurrent exercise prescription guide combined with pharmacological treatment, compared to pharmacological treatment alone, in controlling cardiovascular risk factors and physical capacity in adult users of the Cardiovascular Health Program at the External CESFAM in Valdivia during 2024? Hypothesis H1: The efficacy of a personalized concurrent exercise prescription guide combined with pharmacological treatment is greater than pharmacological treatment alone in controlling cardiovascular risk factors (CVRF) and physical capacity in adult users of the Cardiovascular Health Program at the External CESFAM in Valdivia during 2024. (group difference hypothesis) H0: The efficacy of a personalized concurrent exercise prescription guide combined with pharmacological treatment is equal to pharmacological treatment alone in controlling CVRF and physical capacity in adult users of the Cardiovascular Health Program at the External CESFAM in Valdivia during 2024. (group difference hypothesis) Statistical Hypothesis

Group difference hypothesis:

* H0: μA = μB
* H1: μA > μB OBJECTIVES General Objective To determine the efficacy of a personalized concurrent exercise prescription guide combined with pharmacological treatment, compared to pharmacological treatment alone, in controlling cardiovascular risk factors and physical capacity in adult users of the Cardiovascular Health Program at the External CESFAM in Valdivia during 2024.

2.2.2 Specific Objectives

* To describe the effects of applying a personalized concurrent exercise prescription guide on cardiovascular risk factors in adult users of the Cardiovascular Health Program at the External CESFAM in Valdivia.
* To describe the effects of applying a personalized concurrent exercise prescription guide on physical capacity in adult users of the Cardiovascular Health Program at the External CESFAM in Valdivia.
* To evaluate adherence to the personalized concurrent exercise guide and pharmacological treatment in adult users of the Cardiovascular Health Program at the External CESFAM in Valdivia.
* To describe the clinical significance of the interventions through the calculation of effect size and the clinical relevance perceived by the participants regarding the interventions.

2.3 METHODOLOGY AND PROCEDURES Research Design The research design corresponds to a pilot randomized controlled clinical trial (RCT) with parallel groups and superiority. This design aligns with the general objective and proposed hypothesis, aiming to evaluate the efficacy of a personalized concurrent exercise prescription guide combined with pharmacological treatment, compared to pharmacological treatment alone, in controlling cardiovascular risk factors and physical capacity.

The primary study variables include blood pressure, fasting glucose, total cholesterol, and triglycerides, which are standard measurements for the Cardiovascular Health Program. Secondary variables include sociodemographic and medical background, level of physical activity, muscle strength, cardiorespiratory capacity, body composition, adherence to the exercise guide, and patient perception of changes experienced due to the intervention.

Population The study population will consist of adult users of the Cardiovascular Health Program (PSCV) enrolled in the External CESFAM in Valdivia. The research team will directly invite PSCV users during their regular check-up hours. Research professionals will be properly identified as staff from Universidad San Sebastián and will provide detailed information about the research, the exercise prescription guide application, program duration, benefits, and risks. Interested participants will be asked to sign informed consent. The recruitment period will last up to 1 month, extendable by another month if necessary to obtain the required sample size.

Sample Size Calculation

The sample size calculation is based on recommendations from the literature for pilot studies and includes:

* T-test - Means: difference between two independent means,
* Type I error: 5%,
* Statistical power: 80%,
* Effect size (ES): 0.5 according to Cohen's classification. Using these parameters, the recommended total sample size is fifteen subjects per group. Assuming a 30% dropout rate, the total population will correspond to thirty-nine participants. After the eligibility process, participants will be randomly assigned to an experimental group (EG) and a control group (CG) using a 1:1 allocation ratio through an online randomization system. Allocation concealment will be maintained using opaque, sealed, and consecutively numbered envelopes.

The experimental group will receive the intervention based on the personalized exercise prescription guide plus their usual pharmacological treatment associated with the PSCV, while the control group will maintain their usual pharmacological treatment associated with the PSCV.

Information Production Techniques All evaluations will be performed pre- and post-intervention in both the experimental and control groups.

Clinical Record Review:

The PSCV's responsible physician, with prior authorization from the External CESFAM's management and approval from the Valdivia Health Service Ethics Committee, will review the participants' medical records, collecting information on sociodemographic and medical background: sex, age, education, time in the cardiovascular health program, medical history, medications, dosage, and duration of medication use. These variables will be used to characterize the study sample.

Evaluations and follow-up will be conducted by trained Kinesiologists in evaluation techniques, exercise prescription, and cardiovascular risk factors, at the University of San Sebastián Health Center in Valdivia. A professional Kinesiologist will measure the variables, blinded to the participant's intervention assignment. These evaluations will encompass Cardiovascular Variables Evaluation, Cardiovascular Risk Factor, Metabolic Variables, Health-related Physical Capacity, Adherence to Treatment, and the Global Rating of Change Scale.

2.4 ANALYSIS OF ETHICAL IMPLICATIONS Risk-Benefit Analysis This study adheres to the Declaration of Helsinki, ensuring informed consent is obtained from all participants. The intervention will be conducted in both groups, with evaluations presenting minimal risk. Users may experience post-exercise muscle fatigue, which could last up to 48 hours, mitigated through education about exercise effects. The benefits include updated knowledge about participants' health status and physical capacity, with personalized exercise shown to effectively control cardiovascular risk factors.

Confidentiality Protection The clinical record review will be conducted at the External CESFAM by the PSCV responsible, and physical evaluations will be conducted at the University of San Sebastián Health Center. Participants will be assigned unique codes to preserve anonymity, with informed consent clearly stating data will not be used for purposes other than the study. Collected information will be stored securely by the Principal Investigator for 4 years, after which it will be handed over to the CESFAM. Only the research team will have access to the results.

ELIGIBILITY:
Inclusion Criteria:

1. Being physically inactive (not engaging in 300 or 150 minutes of moderate or vigorous intensity physical activity per week, respectively, as measured by the IPAQ questionnaire);
2. Body mass index between 25 and 39.9 kg/m²;
3. Enrolled in the Cardiovascular Health Program;
4. Diagnosis of hypertension with the use of 1 and/or 2 antihypertensive medications;
5. Diagnosis of Type 2 Diabetes Mellitus with the use of 1 oral hypoglycemic agent, non-insulin-dependent;
6. Diagnosis of dyslipidemia with the use of 1 lipid-lowering agent;
7. Possession of a telephone device.

Exclusion Criteria:

1. Bone disease;
2. Ischemic disease or arrhythmia;
3. Chronic respiratory disease;
4. Uncontrolled chronic diseases;
5. Inability to provide informed consent or comply with the tests and exercise protocol for any reason;
6. History of oncological disease or being under investigation for suspected neoplastic disease in any part of the body;
7. Female participants who are pregnant.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-12-29 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Systolic and Diastolic Blood Pressure | Pre-Intervention: Initial assessment before starting the training program. Post-Intervention (Week 6): Final evaluation after 6 weeks.
  Pressure in the arteries during and between heartbeats. (mmHg)
Mean Arterial Pressure (MAP) | Pre-Intervention: Initial assessment before starting the training program. Post-Intervention (Week 6): Final evaluation after 6 weeks.
  Measure of the average pressure in a person's arteries during one cardiac cycle. MAP=Diastolic Blood Pressure + 1/3 (Systolic Blood Pressure-Diastolic Blood Pressure). mmHg
Heart Rate | Pre-Intervention: Initial assessment before starting the training program. Post-Intervention (Week 6): Final evaluation after 6 weeks.
  Number of heartbeats per minute. (bpm)
Fasting Glucose | Pre-Intervention: Initial assessment before starting the training program. Post-Intervention (Week 6): Final evaluation after 6 weeks.
  Blood glucose level after a fasting period. (mg/dL)
Cholesterol | Pre-Intervention: Initial assessment before starting the training program. Post-Intervention (Week 6): Final evaluation after 6 weeks.
  Blood cholesterol refers to the total amount of cholesterol present in the bloodstream. (mg/dL)
Triglycerides | Pre-Intervention: Initial assessment before starting the training program. Post-Intervention (Week 6): Final evaluation after 6 weeks.
  Blood triglycerides are a type of fat (lipid) found in the bloodstream. (mg/dL)
Body Mass Index | Pre-Intervention: Initial assessment before starting the training program. Post-Intervention (Week 6): Final evaluation after 6 weeks.
  The Body Mass Index (BMI) is a metric used to assess the relationship between an individual's weight and height, thereby estimating their weight category, which can range from underweight to obesity. It is calculated by dividing a person's weight in kilograms by the square of their height in meters.
  The formula is: BMI = weight (kg) / [height (m)]^2
  The unit of measurement for BMI is kg/m² (kilograms per square meter).
Lean Mass | Pre-Intervention: Initial assessment before starting the training program. Post-Intervention (Week 6): Final evaluation after 6 weeks.
  Lean mass, also known as lean body mass, refers to the portion of the body that is not composed of fat. It includes muscles, bones, internal organs, skin, body water, and other fat-free tissues. The unit of measurement for lean mass is (%).
Fat Mass | Pre-Intervention: Initial assessment before starting the training program. Post-Intervention (Week 6): Final evaluation after 6 weeks.
  Fat mass refers to the total amount of fat tissue in the body. The unit of measurement for lean mass is (%).
Handgrip strength | Pre-Intervention: Initial assessment before starting the training program. Post-Intervention (Week 6): Final evaluation after 6 weeks.
  Handgrip Dynamometry: Measurement of handgrip strength. (kgf)
Cardiorespiratory fitness | Pre-Intervention: Initial assessment before starting the training program. Post-Intervention (Week 6): Final evaluation after 6 weeks.
  2-Minute Step Test (2MST): is a functional fitness assessment used to evaluate an individual's cardiorespiratory fitness. During this test, the participant is instructed to march in place for two minutes, lifting their knees to a height midway between the patella (kneecap) and the iliac crest (hip bone). The goal is to count the number of times the right knee reaches the target height within the two-minute period. The primary unit of measurement for the 2-Minute Step Test is the number of steps, specifically the number of times the right knee reaches the required height within the two-minute duration.
VO2 peak | Pre-Intervention: Initial assessment before starting the training program. Post-Intervention (Week 6): Final evaluation after 6 weeks.
  Peak oxygen consumption (VO2peak) refers to the maximum amount of oxygen the body can utilize during intense exercise. It is measured in milliliters of oxygen consumed per kilogram of body weight per minute (ml/kg/min). Using the number of steps in the 2-minute walk test, VO2peak will be estimated. The equation to estimate peak oxygen consumption is: VO2 (mL⋅kg-1⋅min-1) = 13.341 + 0.138 × total steps - (0.183 × BMI).
Treatment Adherence | Post-Intervention (Week 6): Final evaluation after 6 weeks.
  In the context of this study, treatment adherence refers to the extent to which participants follow the prescribed physical exercise regimen. This variable is operationalized as the completion of at least 70% of the scheduled exercise sessions. A participant will be considered "adherent" if they complete at least 70% of the scheduled exercise sessions, according to the data obtained through the described measurement methods. This figure is calculated by dividing the number of completed sessions by the total number of scheduled sessions and multiplying the result by 100.
Global Rating Scale | Pre-Intervention: Initial assessment before starting the training program. Post-Intervention (Week 6): Final evaluation after 6 weeks.
  The Global Rating Scale (GRS) will be applied as an instrument for evaluating the patient's perception of changes experienced in their health status, functionality, or symptoms. The methodology for implementing the GRS will involve asking patients to provide a rating of their current health status compared to an established reference point, which, in our case, will be the beginning of the study.
  The GRS will be presented in two formats: Numeric: Offering a range that can vary, for example, from -7 (much worse) to +7 (much better), allowing for a gradable assessment of changes. Descriptive: Providing qualitative terms such as "much worse," "no change," or "much better," facilitating patients' expression of their perception of change in a more narrative manner.
  The "unit" of measurement for the GRS is the position on the numeric scale or the descriptive term that best represents the patient's perception of change.

SECONDARY OUTCOMES:
Gender | Pre-Intervention: Initial assessment before starting the training program.
  Gender: Biological classification of the individual. (No unit of measure)
Age | Pre-Intervention: Initial assessment before starting the training program.
  Age: Number of complete years since birth. (Years)
Ancestry | Pre-Intervention: Initial assessment before starting the training program.
  Ancestry: Ethnic or racial origin of the individual. (No unit of measure)
Education Level | Pre-Intervention: Initial assessment before starting the training program.
  Education Level: Highest level of education achieved. (No unit of measure)
Duration in Cardiovascular Health Program | Pre-Intervention: Initial assessment before starting the training program.
  Duration in Cardiovascular Health Program: Length of participation in the program. (Months or Years)
Morbid Background | Pre-Intervention: Initial assessment before starting the training program.
  Morbid Background: History of previous diseases and medical conditions. (No unit of measure)
Medications and Dosage: | Pre-Intervention: Initial assessment before starting the training program.
  Medications and Dosage: Description of used medications and their dosages. (mg/day or as prescribed)
Duration of Medication Use | Pre-Intervention: Initial assessment before starting the training program.
  Duration of Medication Use: Length of time medications have been used. (Months or Years)
Physical Activity Level | Pre-Intervention: Initial assessment before starting the training program.
  The International Physical Activity Questionnaire (IPAQ) is a recognized instrument for assessing physical activity in adults. This survey outlines the frequency (measured in days per week) and duration (hours and minutes per day) of physical activities categorized into four intensity levels: sedentary, walking, moderate physical activity, and vigorous physical activity.
  For each intensity level, the units of measurement are expressed in days per week and hours or minutes per day, with specific Metabolic Equivalent Task (METs) values assigned to each activity (Walking: 3.3 METs, Moderate Physical Activity: 4 METs, Vigorous Physical Activity: 8 METs). The responses can be converted into MET-minutes/week, enabling a quantitative and consistent comparison of total physical activity, encompassing various types and intensities.
Height | Pre-Intervention: Initial assessment before starting the training program.
  Individual's height. (cm)
Weight | Pre-Intervention: Initial assessment before starting the training program. Post-Intervention (Week 6): Final evaluation after 6 weeks.
  Total body mass. (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Johnattan Cano Montoya, MSc., Study Chair — Universidad San Sebastián; Johnattan Cano Montoya, MSc., Study Director — Universidad San Sebastián; Johnattan Cano Montoya, MSc., Principal Investigator — Universidad San Sebastián
Locations (1):
- Universidad San Sebastián, Valdivia, Los Ríos Region, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yusuf S, Joseph P, Rangarajan S, Islam S, Mente A, Hystad P, Brauer M, Kutty VR, Gupta R, Wielgosz A, AlHabib KF, Dans A, Lopez-Jaramillo P, Avezum A, Lanas F, Oguz A, Kruger IM, Diaz R, Yusoff K, Mony P, Chifamba J, Yeates K, Kelishadi R, Yusufali A, Khatib R, Rahman O, Zatonska K, Iqbal R, Wei L, Bo H, Rosengren A, Kaur M, Mohan V, Lear SA, Teo KK, Leong D, O'Donnell M, McKee M, Dagenais G. Modifiable risk factors, cardiovascular disease, and mortality in 155 722 individuals from 21 high-income, middle-income, and low-income countries (PURE): a prospective cohort study. Lancet. 2020 Mar 7;395(10226):795-808. doi: 10.1016/S0140-6736(19)32008-2. Epub 2019 Sep 3. PMID 31492503
- [Background] Nazzal C, Lefian A, Alonso F. [Incidence of acute myocardial infarction in Chile between 2008 and 2016]. Rev Med Chil. 2021 Mar;149(3):323-329. doi: 10.4067/s0034-98872021000300323. Spanish. PMID 34479310
- [Background] Parra-Soto S, Petermann-Rocha F, Martinez-Sanguinetti MA, Leiva-Ordenez AM, Troncoso-Pantoja C, Ulloa N, Diaz-Martinez X, Celis-Morales C. [Cancer in Chile and worldwide: an overview of the current and future epidemiological context]. Rev Med Chil. 2020 Oct;148(10):1489-1495. doi: 10.4067/S0034-98872020001001489. Spanish. PMID 33844720
- [Background] Celis-Morales C, Salas C, Martinez MA, Leiva AM, Garrido-Mendez A, Diaz-Martinez X. [The economic burden of physical inactivity in Chile]. Rev Med Chil. 2017 Aug;145(8):1091-1092. doi: 10.4067/s0034-98872017000801091. No abstract available. Spanish. PMID 29189871
- [Background] Pratt M, Macera CA, Wang G. Higher direct medical costs associated with physical inactivity. Phys Sportsmed. 2000 Oct;28(10):63-70. doi: 10.3810/psm.2000.10.1237. PMID 20086598
- [Background] Teo KK, Rafiq T. Cardiovascular Risk Factors and Prevention: A Perspective From Developing Countries. Can J Cardiol. 2021 May;37(5):733-743. doi: 10.1016/j.cjca.2021.02.009. Epub 2021 Feb 19. PMID 33610690
- [Background] Pucci GC, Rech CR, Fermino RC, Reis RS. Association between physical activity and quality of life in adults. Rev Saude Publica. 2012 Feb;46(1):166-79. doi: 10.1590/s0034-89102012000100021. English, Portuguese. PMID 22249758
- [Background] Geidl W, Schlesinger S, Mino E, Miranda L, Pfeifer K. Dose-response relationship between physical activity and mortality in adults with noncommunicable diseases: a systematic review and meta-analysis of prospective observational studies. Int J Behav Nutr Phys Act. 2020 Aug 26;17(1):109. doi: 10.1186/s12966-020-01007-5. PMID 32843054
- [Background] DeMarco VG, Aroor AR, Sowers JR. The pathophysiology of hypertension in patients with obesity. Nat Rev Endocrinol. 2014 Jun;10(6):364-76. doi: 10.1038/nrendo.2014.44. Epub 2014 Apr 15. PMID 24732974
- [Background] Bergouignan A, Rudwill F, Simon C, Blanc S. Physical inactivity as the culprit of metabolic inflexibility: evidence from bed-rest studies. J Appl Physiol (1985). 2011 Oct;111(4):1201-10. doi: 10.1152/japplphysiol.00698.2011. Epub 2011 Aug 11. PMID 21836047
- [Background] Yusuf S, Hawken S, Ounpuu S, Dans T, Avezum A, Lanas F, McQueen M, Budaj A, Pais P, Varigos J, Lisheng L; INTERHEART Study Investigators. Effect of potentially modifiable risk factors associated with myocardial infarction in 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):937-52. doi: 10.1016/S0140-6736(04)17018-9. PMID 15364185
- [Background] Diaz-Martinez X, Petermann F, Leiva AM, Garrido-Mendez A, Salas-Bravo C, Martinez MA, Labrana AM, Duran E, Valdivia-Moral P, Zagalaz ML, Poblete-Valderrama F, Alvarez C, Celis-Morales C. [Association of physical inactivity with obesity, diabetes, hypertension and metabolic syndrome in the chilean population]. Rev Med Chil. 2018 May;146(5):585-595. doi: 10.4067/s0034-98872018000500585. Spanish. PMID 30148922
- [Background] Lear SA, Hu W, Rangarajan S, Gasevic D, Leong D, Iqbal R, Casanova A, Swaminathan S, Anjana RM, Kumar R, Rosengren A, Wei L, Yang W, Chuangshi W, Huaxing L, Nair S, Diaz R, Swidon H, Gupta R, Mohammadifard N, Lopez-Jaramillo P, Oguz A, Zatonska K, Seron P, Avezum A, Poirier P, Teo K, Yusuf S. The effect of physical activity on mortality and cardiovascular disease in 130 000 people from 17 high-income, middle-income, and low-income countries: the PURE study. Lancet. 2017 Dec 16;390(10113):2643-2654. doi: 10.1016/S0140-6736(17)31634-3. Epub 2017 Sep 21. PMID 28943267
- [Background] Cristi-Montero C, Ramirez-Campillo R, Alvarez C, Garrido Mendez A, Martinez MA, Diaz Martinez X, Leiva AM, Salas C, Gutierrez M, Sanzana-Inzunza R, Duran E, Labrana AM, Aguilar-Farias N, Celis-Morales C. [Inverse association of cardiorespiratory fitness with cardiovascular risk factors in Chilean adults]. Rev Med Chil. 2016 Aug;144(8):980-989. doi: 10.4067/S0034-98872016000800004. Spanish. PMID 27905643
- [Background] Arija V, Villalobos F, Pedret R, Vinuesa A, Timon M, Basora T, Aguas D, Basora J; Pas-a-Pas research group. Effectiveness of a physical activity program on cardiovascular disease risk in adult primary health-care users: the "Pas-a-Pas" community intervention trial. BMC Public Health. 2017 Jun 15;17(1):576. doi: 10.1186/s12889-017-4485-3. PMID 28619115
- [Background] Pavey TG, Taylor AH, Fox KR, Hillsdon M, Anokye N, Campbell JL, Foster C, Green C, Moxham T, Mutrie N, Searle J, Trueman P, Taylor RS. Effect of exercise referral schemes in primary care on physical activity and improving health outcomes: systematic review and meta-analysis. BMJ. 2011 Nov 4;343:d6462. doi: 10.1136/bmj.d6462. PMID 22058134
- [Background] Campbell F, Holmes M, Everson-Hock E, Davis S, Buckley Woods H, Anokye N, Tappenden P, Kaltenthaler E. A systematic review and economic evaluation of exercise referral schemes in primary care: a short report. Health Technol Assess. 2015 Jul;19(60):1-110. doi: 10.3310/hta19600. PMID 26222987
- [Background] Williams NH, Hendry M, France B, Lewis R, Wilkinson C. Effectiveness of exercise-referral schemes to promote physical activity in adults: systematic review. Br J Gen Pract. 2007 Dec;57(545):979-86. doi: 10.3399/096016407782604866. PMID 18252074
- [Background] Cano-Montoya J, Ramirez-Campillo R, Sade Calles F, Izquierdo M, Fritz Silva N, Arteaga San Martin R, Alvarez C. [Effects of a six weeks exercise training program for type 2 diabetes mellitus and hypertensive patients]. Rev Med Chil. 2018 Jun;146(6):693-701. doi: 10.4067/s0034-98872018000600693. Spanish. PMID 30148900
- [Background] Cano-Montoya J, Ramirez-Campillo R, Martinez C, Sade-Calles F, Salas-Parada A, Alvarez C. [Interaction between antihypertensive therapy and exercise training therapy requires drug regulation in hypertensive patients]. Rev Med Chil. 2016 Feb;144(2):152-61. doi: 10.4067/S0034-98872016000200002. Spanish. PMID 27092668
- [Background] Alvarez C, Ramirez-Campillo R, Martinez-Salazar C, Mancilla R, Flores-Opazo M, Cano-Montoya J, Ciolac EG. Low-Volume High-Intensity Interval Training as a Therapy for Type 2 Diabetes. Int J Sports Med. 2016 Aug;37(9):723-9. doi: 10.1055/s-0042-104935. Epub 2016 Jun 3. PMID 27259099
- [Background] Cadore EL, Izquierdo M. How to simultaneously optimize muscle strength, power, functional capacity, and cardiovascular gains in the elderly: an update. Age (Dordr). 2013 Dec;35(6):2329-44. doi: 10.1007/s11357-012-9503-x. Epub 2013 Jan 4. PMID 23288690
- [Background] Teodoro JL, Izquierdo M, da Silva LXN, Baroni BM, Grazioli R, Lopez P, Fritsch CG, Radaelli R, Saez de Asteasu ML, Bottaro M, Farinha JB, Pinto RS, Cadore EL. Effects of long-term concurrent training to failure or not in muscle power output, muscle quality and cardiometabolic risk factors in older men: A secondary analysis of a randomized clinical trial. Exp Gerontol. 2020 Oct 1;139:111023. doi: 10.1016/j.exger.2020.111023. Epub 2020 Jul 19. PMID 32697957
- [Background] Higham SM, Mendham AE, Rosenbaum S, Allen NG, Smith G, Stadnyk A, Duffield R. Effects of concurrent exercise training on body composition, systemic inflammation, and components of metabolic syndrome in inactive academics: a randomised controlled trial. Eur J Appl Physiol. 2023 Apr;123(4):809-820. doi: 10.1007/s00421-022-05108-w. Epub 2022 Dec 6. PMID 36471186
- [Background] Alvarez C, Ramirez-Velez R, Ramirez-Campillo R, Lucia A, Alonso-Martinez AM, Faundez H, Cadore EL, Izquierdo M. Improvements cardiometabolic risk factors in Latin American Amerindians (the Mapuche) with concurrent training. Scand J Med Sci Sports. 2019 Jun;29(6):886-896. doi: 10.1111/sms.13409. Epub 2019 Mar 12. PMID 30770586
- [Background] Amaro-Gahete FJ, Ponce-Gonzalez JG, Corral-Perez J, Velazquez-Diaz D, Lavie CJ, Jimenez-Pavon D. Effect of a 12-Week Concurrent Training Intervention on Cardiometabolic Health in Obese Men: A Pilot Study. Front Physiol. 2021 Feb 11;12:630831. doi: 10.3389/fphys.2021.630831. eCollection 2021. PMID 33643072
- [Background] Gao J, Yu L. Effects of concurrent training sequence on VO2max and lower limb strength performance: A systematic review and meta-analysis. Front Physiol. 2023 Jan 26;14:1072679. doi: 10.3389/fphys.2023.1072679. eCollection 2023. PMID 36776981
- [Background] Gibala MJ, Little JP, Macdonald MJ, Hawley JA. Physiological adaptations to low-volume, high-intensity interval training in health and disease. J Physiol. 2012 Mar 1;590(5):1077-84. doi: 10.1113/jphysiol.2011.224725. Epub 2012 Jan 30. PMID 22289907
- [Background] Hawley JA, Hargreaves M, Joyner MJ, Zierath JR. Integrative biology of exercise. Cell. 2014 Nov 6;159(4):738-49. doi: 10.1016/j.cell.2014.10.029. PMID 25417152
- [Background] Coffey VG, Hawley JA. The molecular bases of training adaptation. Sports Med. 2007;37(9):737-63. doi: 10.2165/00007256-200737090-00001. PMID 17722947
- [Background] Goodpaster BH, Sparks LM. Metabolic Flexibility in Health and Disease. Cell Metab. 2017 May 2;25(5):1027-1036. doi: 10.1016/j.cmet.2017.04.015. PMID 28467922
- [Background] Freese J, Klement RJ, Ruiz-Nunez B, Schwarz S, Lotzerich H. The sedentary (r)evolution: Have we lost our metabolic flexibility? F1000Res. 2017 Oct 2;6:1787. doi: 10.12688/f1000research.12724.2. eCollection 2017. PMID 29225776
- [Background] Pedersen BK, Saltin B. Exercise as medicine - evidence for prescribing exercise as therapy in 26 different chronic diseases. Scand J Med Sci Sports. 2015 Dec;25 Suppl 3:1-72. doi: 10.1111/sms.12581. PMID 26606383
- [Background] Islam H, Gibala MJ, Little JP. Exercise Snacks: A Novel Strategy to Improve Cardiometabolic Health. Exerc Sport Sci Rev. 2022 Jan 1;50(1):31-37. doi: 10.1249/JES.0000000000000275. PMID 34669625
- [Background] Thornton JS, Fremont P, Khan K, Poirier P, Fowles J, Wells GD, Frankovich RJ. Physical activity prescription: a critical opportunity to address a modifiable risk factor for the prevention and management of chronic disease: a position statement by the Canadian Academy of Sport and Exercise Medicine. Br J Sports Med. 2016 Sep;50(18):1109-14. doi: 10.1136/bjsports-2016-096291. Epub 2016 Jun 22. PMID 27335208
- [Background] Moore CG, Carter RE, Nietert PJ, Stewart PW. Recommendations for planning pilot studies in clinical and translational research. Clin Transl Sci. 2011 Oct;4(5):332-7. doi: 10.1111/j.1752-8062.2011.00347.x. PMID 22029804
- [Background] Christensen E. Methodology of superiority vs. equivalence trials and non-inferiority trials. J Hepatol. 2007 May;46(5):947-54. doi: 10.1016/j.jhep.2007.02.015. Epub 2007 Mar 9. PMID 17412447
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Takahashi H, Yoshika M, Yokoi T. Validation of three automatic devices for the self-measurement of blood pressure according to the European Society of Hypertension International Protocol revision 2010: the Omron HEM-7130, HEM-7320F, and HEM-7500F. Blood Press Monit. 2015 Apr;20(2):92-7. doi: 10.1097/MBP.0000000000000096. PMID 25462531
- [Background] Pleus S, Baumstark A, Schauer S, Kolle J, Jendrike N, Mende J, Haug C, Freckmann G. User Performance Evaluation and System Accuracy Assessment of Four Blood Glucose Monitoring Systems With Color Coding of Measurement Results. J Diabetes Sci Technol. 2024 May;18(3):644-652. doi: 10.1177/19322968221141926. Epub 2022 Nov 26. PMID 36433806
- [Background] Coqueiro Rda S, Santos MC, Neto Jde S, Queiroz BM, Brugger NA, Barbosa AR. Validity of a portable glucose, total cholesterol, and triglycerides multi-analyzer in adults. Biol Res Nurs. 2014 Jul;16(3):288-94. doi: 10.1177/1099800413495953. Epub 2013 Jul 19. PMID 23871994
- [Background] Huang L, Liu Y, Lin T, Hou L, Song Q, Ge N, Yue J. Reliability and validity of two hand dynamometers when used by community-dwelling adults aged over 50 years. BMC Geriatr. 2022 Jul 15;22(1):580. doi: 10.1186/s12877-022-03270-6. PMID 35840905
- [Background] Geeta A, Jamaiyah H, Safiza MN, Khor GL, Kee CC, Ahmad AZ, Suzana S, Rahmah R, Faudzi A. Reliability, technical error of measurements and validity of instruments for nutritional status assessment of adults in Malaysia. Singapore Med J. 2009 Oct;50(10):1013-8. PMID 19907894
- [Background] Vasold KL, Parks AC, Phelan DML, Pontifex MB, Pivarnik JM. Reliability and Validity of Commercially Available Low-Cost Bioelectrical Impedance Analysis. Int J Sport Nutr Exerc Metab. 2019 Jul 1;29(4):406-410. doi: 10.1123/ijsnem.2018-0283. PMID 30507268
- [Background] Guyatt GH, Osoba D, Wu AW, Wyrwich KW, Norman GR; Clinical Significance Consensus Meeting Group. Methods to explain the clinical significance of health status measures. Mayo Clin Proc. 2002 Apr;77(4):371-83. doi: 10.4065/77.4.371. PMID 11936935
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Alvarez C, Ramirez-Campillo R, Lucia A, Ramirez-Velez R, Izquierdo M. Concurrent exercise training on hyperglycemia and comorbidities associated: Non-responders using clinical cutoff points. Scand J Med Sci Sports. 2019 Jul;29(7):952-967. doi: 10.1111/sms.13413. Epub 2019 Apr 9. PMID 30825342
- [Background] Ciolac EG, Mantuani SS, Neiva CM, Verardi C, Pessoa-Filho DM, Pimenta L. Rating of perceived exertion as a tool for prescribing and self regulating interval training: a pilot study. Biol Sport. 2015 Jun;32(2):103-8. doi: 10.5604/20831862.1134312. Epub 2015 Jan 15. PMID 26028809
- [Background] Robertson RJ, Goss FL, Rutkowski J, Lenz B, Dixon C, Timmer J, Frazee K, Dube J, Andreacci J. Concurrent validation of the OMNI perceived exertion scale for resistance exercise. Med Sci Sports Exerc. 2003 Feb;35(2):333-41. doi: 10.1249/01.MSS.0000048831.15016.2A. PMID 12569225
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT06509282/Prot_SAP_ICF_000.pdf